CLINICAL TRIAL: NCT02855827
Title: Constitution of a Cohort for Monitoring Patients Candidating for Ovarian Tissue Autograft
Acronym: PERIDATOR
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: CHU de Reims (Other); University Hospital, Marseille (Other); University Hospital, Lille (Other); Central Hospital, Nancy, France (Other); University Hospital, Grenoble (Other); CMCO SIHCUS, Schiltingheim (Other); University Hospital, Bordeaux (Other); Nantes University Hospital (Other); University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: P/2013/170
Record Dates: First submitted 2016-07-20; First posted 2016-08-04 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-06

CONDITIONS: Ovarian Function Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Ovarian cryopreservation is one of the available option for preserving fertility prior to potentially sterilizing treatments. In the absence of other techniques such as in vitro folliculogenesis or injection of isolated ovarian follicles, this tissue can only be re-used by autograft. In France, the first live birth after orthotopic ovarian transplantation, was obtained by Roux et al. in 2009.

This clinical trial aims to build a cohort of patients likely to use their ovarian tissue cryopreserved by autograft.

DETAILED DESCRIPTION:
Ovarian cryopreservation is one of the available option for preserving fertility prior to potentially sterilizing treatments. In the absence of other techniques such as in vitro folliculogenesis or injection of isolated ovarian follicles, this tissue can only be re-used by autograft. In France, the first live birth after orthotopic ovarian transplantation, was obtained by Roux et al. in 2009.

This clinical trial aims to build a cohort of patients likely to use their ovarian tissue cryopreserved by autograft. This cohort will be used to:

* Follow up of patients with their cryopreserved ovarian tissue;
* Evaluate requests for ovarian tissue grafting ;
* Propose a search of residual disease in case of neoplastic disease risk (if possible);
* Allowing patients to benefit from an ovarian tissue autograft;
* Assess the effectiveness of autograft technique after the restoration of ovarian function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have cryopreserved their ovarian tissue;
* Patients with premature ovarian insufficiency;
* Patients older than 11 years (bone age) for induction of puberty;
* Patients aged from 18 to 43 years for the restoration of ovarian function;
* No objection from the patient
* Patients who have already received ovarian tissue autograft.

Exclusion Criteria:

* Patients aged under 11 years (bone age);
* Patients older than 43 years;
* Patients refusing to be included;
* Patients (adults) under guardianship, curators and safeguard justice

Ages: 11 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients likely to re-use their ovarian tissue cryopreserved by autograft
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2013-05 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Number of patient who are candidate to ovarian tissue autograft | 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Besancon, Besançon, France

REFERENCES:
- [Background] Roux C, Amiot C, Agnani G, Aubard Y, Rohrlich PS, Piver P. Live birth after ovarian tissue autograft in a patient with sickle cell disease treated by allogeneic bone marrow transplantation. Fertil Steril. 2010 May 1;93(7):2413.e15-9. doi: 10.1016/j.fertnstert.2009.12.022. Epub 2010 Feb 1. PMID 20117783
- [Background] Amiot C, Angelot-Delettre F, Zver T, Alvergnas-Vieille M, Saas P, Garnache-Ottou F, Roux C. Minimal residual disease detection of leukemic cells in ovarian cortex by eight-color flow cytometry. Hum Reprod. 2013 Aug;28(8):2157-67. doi: 10.1093/humrep/det126. Epub 2013 Apr 30. PMID 23633552
- [Background] Fauque P, Ben Amor A, Joanne C, Agnani G, Bresson JL, Roux C. Use of trypan blue staining to assess the quality of ovarian cryopreservation. Fertil Steril. 2007 May;87(5):1200-7. doi: 10.1016/j.fertnstert.2006.08.115. Epub 2007 Feb 20. PMID 17307173